CLINICAL TRIAL: NCT06367257
Title: App-based Recording and Optimization of the Nutritional Status in Patients With Head and Neck Tumors During and After Radio(Chemo)Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Emento App
Record Dates: First submitted 2024-04-03; First posted 2024-04-16 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Squamous Cell Carcinoma of Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- App Usage (Experimental): Patients receive the daily reminder message via app (Emento) that they should pay attention to sufficient calorie intake. In addition, these patients receive 3 screening questions about their current health and nutritional status twice a week.
  Interventions: Procedure: App Usage
- Standard (Other): Patients in the control arm receive supportive care during and after radio(chemo)therapy according to hospital standards.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Procedure: App Usage — Conducting patient surveys with app
  Arms: App Usage
Other: Standard of Care — supportive care during and after radio(chemo)therapy according to hospial standards
  Arms: Standard

SUMMARY:
Patients with head and neck cancer requiring definitive or adjuvant radio(chemo)therapy can take part in the study. The aim is to record the nutritional status and diet of the patients during the trial and regularly at a period of 8 weeks after irradiation and to reduce the rate of weight loss and malnutrition.

DETAILED DESCRIPTION:
Patients with head and neck cancer requiring definitive or adjuvant radio(chemo)therapy can take part in the study. The aim is to record the nutritional status and diet of the patients during the trial and regularly at a period of 8 weeks after irradiation and to reduce the rate of weight loss and malnutrition.

Patients in the experimental arm receive the daily reminder message via app (Emento) that they should pay attention to adequate caloric intake. In addition, these patients receive 3 screening questions about their current health and nutritional status twice a week.

In case of relevant deterioration (any negative value in the screening questions is explained under study procedure), additional further questions are asked, which are specifically aimed at the side effects of the tumor therapy (mainly dysphagia, pain). The answers will be transmitted to the radiation clinic.

If a question is answered positively, this is reported to the radiotherapy clinic on the one hand and on the other hand, the patient is asked to consult the doctor in the clinic as soon as possible.

ELIGIBILITY:
Inclusion Criteria:

* Patients with squamous cell carcinoma in the head and neck region, who receive a postsurgical or definitive radio(chemo)therapy
* Patients who have a smartphone on which the Emento app can be installed
* Minimum age 18 years

Exclusion Criteria:

* Patients who are represented by a legal guardian
* Patients who are not suitable for participation in the study due to a language barrier

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2024-02-29 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in rates of weight loss with additional app-based Patient Care | during trial, about 24 months

SECONDARY OUTCOMES:
Frequency of deteriorations in health status subjectively reported by patients and recorded via the app. | during trial, about 24 months
Frequency of additional app-triggered contacts of the clinic with the patients | during trial, about 24 months
Frequency of critical health conditions (physician-verified) detected earlier by the app. | during trial, about 24 months
Change in quality of life measured per questionnaires | during trial, about 24 months
Change of incidence of malnutrition and sarcopenia before, during and after radio(chemo)therapy. | during trial, about 24 months
Change of course of malnutrition and sarcopenia before, during and after radio(chemo)therapy. | during trial, about 24 months
Rate of therapy interruptions/discontinuations | during trial, about 24 months
Overall survival | during trial, about 24 months
Disease-free/progression-free survival | during trial, about 24 months
Change of Loco-regional tumor control | during trial, about 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Marlen Haderlein, PD, Study Director — Universitätsklinikum Erlangen, Radiation Oncology; Luitpold Distel, Prof., Study Director — Universitätsklinikum Erlangen, Radiation Oncology; Allison Lamrani, Principal Investigator — Universitätsklinikum Erlangen, Radiation Oncology; Charlotte Schmitter, Dr., Principal Investigator — Universitätsklinikum Erlangen, Radiation Oncology
Locations (1):
- Universitätsklinikum Erlangen, Strahlenklinik, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No